CLINICAL TRIAL: NCT03257137
Title: Diet and Sleep Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 17-0616
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Diet Modification
Keywords: sleep; macronutrients; dietary patterns; sleep quality; diet quality; polysomnography; appetite; mood; hunger
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will undergo both diet pattern conditions but not be informed of their differences. The technologist scoring the sleep studies and actiwatches will be blinded to the condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Diet (Experimental): This dietary pattern will represent recommendations for fiber and added sugar set forth in the 2015 Dietary Guidelines for Americans and saturated fat guidelines from the American Heart Association
  Interventions: Other: Diet Quality
- Simulated Fast Food (SFF) (Experimental): This dietary pattern will represent the typical American diet for fiber, added sugar, and saturated fat intake.
  Interventions: Other: Diet Quality

INTERVENTIONS:
Other: Diet Quality — Diets matched for calorie intake and macronutrient distribution but differing by overall diet quality will be provided in a random order, cross-over design study.

SUMMARY:
This study will investigate the effect of two dietary patterns on sleep outcomes and measures of reported appetite. Participants will be given two different diets on two separate stays.

DETAILED DESCRIPTION:
Normal sleep consists of alternating periods of non-rapid eye movement (NREM) and rapid eye movement (REM) sleep. The deeper stages of NREM sleep are also known as slow-wave sleep (SWS). Genetic and environmental factors, such as age, gender, race, socioeconomic status and others contribute to high inter-individual variability in sleep quality.

Current evidence from epidemiologic, clinical and experimental studies support a strong relationship between insufficient sleep and increased risk for obesity. A reciprocal connection between sleep and energy metabolism may exist between diet and sleep.

It is also well known that diet greatly influences body weight and metabolic health. Numerous disease risk factors are known to be associated with dietary patters consisting low fiber, high saturated fat, and added sugar, but the effects of diet on sleep quality remains unknown.

A small group of studies have indicated an effect of diet on sleep quality (assessed objectively by polysomnography [PSG]) under controlled laboratory conditions. However, none have experimentally tested sleep and appetite outcomes under different dietary patterns matched for macronutrients.

The overall objective of this study is to compare the effects of consumption of unhealthy meals with low fiber, high saturated fat, and high added sugar content i.e. simulated fast food diet [SFF] to healthy meals with high fiber, low saturated fat, and low added sugar content i.e. healthy diet. We hypothesize that a healthy diet (as recommended by the Dietary Guidelines Advisory Committee and the American Heart Association) compared to SFF diet will promote better sleep quality (as assessed by PSG) reflected by higher sleep efficiency, increased SWS and increased REM sleep and other improved sleep variables. We will also evaluate subjective appetite, mood and sleepiness as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants (age: 21-40 years and BMI=19.0-26.0 kg/m2) who habitually sleep on average 7-8 hours per night (as confirmed by actigraphy) and eat at least 3 meals per day (as confirmed by food diaries) will be studied. Subjects will be required to have stable sleep habits for the past 6 months and stable dietary habits for the past 3 months.

Exclusion Criteria:

* Obstructive sleep apnea by laboratory polysomnography or history of any other sleep disorder, night or rotating shift work (current or in the past 1 year), habitual daytime naps, recent (< 4 week) travel across time zones, extreme chronotypes, any acute or chronic medical condition, prediabetes or diabetes, prior or current eating or psychiatric disorders, claustrophobia, irregular menstrual periods, menopause, currently pregnant (screened with urine test), recently postpartum (within 1 year), currently lactating, alcohol abuse, excessive caffeine intake, smoking, illegal drug use, currently following a weight loss regimen or any other special diet or exercise programs, extreme food allergies or intolerances, and abnormal findings on screening blood testing. Participants will also be required not to take any prescription or over the counter medications, supplements that can affect sleep, metabolism, mood or appetite. Women will be required to not be on hormone replacement therapy.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Sleep quality night 2 | Bedtime (11:00PM) to Wake time (7:30AM)
  Night 2 PSG recordings

SECONDARY OUTCOMES:
Subjective appetite area under the curve | 7:30am-11:00PM
  A collection of all subjective ratings (upon waking, pre and post meals, and hourly)
Subjective appetite daily average | 7:30am-11:00PM
  A collection of all subjective ratings (upon waking, pre and post meals, and hourly)
Mood area under the curve | 7:30am-11:00PM
  A collection of all subjective ratings (upon waking, pre and post meals, and hourly)
Mood daily average | 7:30am-11:00PM
  A collection of all subjective ratings (upon waking, pre and post meals, and hourly)
Subjective sleep quality area under the curve | 7:30am-11:00PM
  A collection of all subjective ratings (upon waking, pre and post meals, and hourly)
Subjective sleep quality daily average | 7:30am-11:00PM
  A collection of all subjective ratings (upon waking, pre and post meals, and hourly)
Sleep quality night 1 | 11:00PM to 7:30AM
  Night 2 PSG recordings
Sleep night 1 | 11:00PM to 7:30AM
  Measured with wrist actigraphy
Sleep night 2 | 11:00PM to 7:30AM
  Measured with wrist actigraphy
Sleep night 3 | 11:00PM to 7:30AM
  Measured with wrist actigraphy

OTHER OUTCOMES:
Appetite upon waking | First response in the morning
  First response in the morning using subjective questionnaires
Mood upon waking | 7:30AM
  First response in the morning using subjective questionnaires
Sleepiness upon waking | 7:30AM
  First response in the morning using subjective questionnaires
Morning appetite | 7:30AM to 11:00AM
  Morning hourly and pre and post meal response using subjective questionnaires
Morning mood | 7:30AM to 11:00AM
  Morning hourly and pre and post meal response using subjective questionnaires
Morning sleepiness | 7:30AM to 11:00AM
  Morning hourly and pre and post meal response using subjective questionnaires
Mid-day appetite | 11:00AM to 5:00PM
  Mid-day hourly and pre and post meal response using subjective questionnaires
Mid-day mood | 11:00AM to 5:00PM
  Mid-day hourly and pre and post meal response using subjective questionnaires
Mid-day sleepiness | 11:00AM to 5:00PM
  Mid-day hourly and pre and post meal response using subjective questionnaires
Evening appetite | 5:00PM to 11:00PM
  Evening hourly and pre and post meal response using subjective questionnaires
Evening mood | 5:00PM to 11:00PM
  Evening hourly and pre and post meal response using subjective questionnaires
Evening sleepiness | 5:00PM to 11:00PM
  Evening hourly and pre and post meal response using subjective questionnaires
Bedtime appetite | Response at bedtime
  Response at bedtime using subjective questionnaires
Bedtime mood | 11:00PM
  Response at bedtime using subjective questionnaires
Bedtime sleepiness | 11:00PM
  Response at bedtime using subjective questionnaires
Average sleep duration | 21 days
  At home wrist actigraphy
Average sleep onset latency | 21 days
  At home wrist actigraphy
Average night-time awakenings | 21 days
  At home wrist actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- Univeristy of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boege HL, Wilson KD, Kilkus JM, Qiu W, Cheng B, Wroblewski KE, Tucker B, Tasali E, St-Onge MP. Higher daytime intake of fruits and vegetables predicts less disrupted nighttime sleep in younger adults. Sleep Health. 2025 Oct;11(5):590-596. doi: 10.1016/j.sleh.2025.05.003. Epub 2025 Jun 11. PMID 40506285